CLINICAL TRIAL: NCT01853475
Title: Open Label, Parallel Group Study to Investigate the Pharmacokinetics (PK) Following Oral Co-administration of Piperaquine Phosphate (PQP) Tablets With a Prototype OZ439 + TPGS Formulation in the Fasted State in Healthy Volunteers
Brief Title: Healthy Volunteer Study of the Pharmacokinetics of Oral Piperaquine With OZ439 + TPGS Formulation in the Fasted State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Richmond Pharmacology Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMV_OZ439_13_002; 2013-000983-28 (EudraCT Number)
Record Dates: First submitted 2013-05-10; First posted 2013-05-15 (Estimated); Results first posted 2015-04-08 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Malaria
Keywords: pharmacokinetics; safety; tolerability; bioavailability
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): PQP tablets 1440mg and OZ439+TPGS 800mg co-administered as a single oral dose fasted.
  Interventions: Drug: PQP tablets 1440mg; Drug: OZ439+TPGS 800mg
- Treatment B (Experimental): PQP tablets 960mg and OZ439+TPGS 800mg co-administered as a single oral dose fasted.
  Interventions: Drug: PQP tablets 960mg; Drug: OZ439+TPGS 800mg
- Treatment C - Reference (Active Comparator): PQP Tablets 1440 mg and OZ439 PIB 800mg + full fat cow's milk
  Interventions: Drug: PQP tablets 1440mg; Drug: OZ439 PIB 800mg

INTERVENTIONS:
Drug: PQP tablets 960mg — Piperaquine phosphate tablets 960mg
  Arms: Treatment B
Drug: PQP tablets 1440mg — Piperaquine phosphate tablets 1440mg
  Arms: Treatment A; Treatment C - Reference
Drug: OZ439+TPGS 800mg — OZ439+TPGS prototype formulation 800mg
  Arms: Treatment A; Treatment B
Drug: OZ439 PIB 800mg — OZ439 Powder in Bottle Aqueous Solution 800mg
  Arms: Treatment C - Reference

SUMMARY:
Piperaquine tablets (coated) + OZ439 granules + TPGS granules will be co-administered in Phase IIb (adults). However, safety and PK data (for OZ439 plus piperaquine) were obtained using piperaquine tablets plus OZ439 as Powder in Bottle with milk. Piperaquine has not yet been administered together with TPGS. Co-administration of piperaquine plus OZ439 as Powder in Bottle (PIB) with milk results in an increase in OZ439 exposure (current estimate ~ 70% due to a small drug drug interaction).

This study investigates the exposure of piperaquine and OZ439 when co-administered as piperaquine phosphate tablets and OZ439 + TPGS prototype (a formulation close to that of Phase IIb, but not identical), in order to select the appropriate doses for Phase IIb. The reference treatment is piperaquine phosphate tablets + OZ439 Powder in Bottle + full fat milk

DETAILED DESCRIPTION:
Objectives:

1. To evaluate the piperaquine and OZ439 pharmacokinetics when administered as a combination of piperaquine phosphate tablets with OZ439 / TPGS formulation in the fasted state
2. To evaluate the piperaquine and OZ439 pharmacokinetics of a reference free combination formulation: piperaquine phosphate tablets with OZ439 powder in bottle (PIB) given with full fat milk
3. To determine safety and tolerability of OZ439 and piperaquine phosphate when co-administered.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male/female of any race aged 18-55 years at screening
2. Body Mass Index 18-30kg/m2; body weight >50kg but no more than 100kg at screening
3. Females with negative pregnancy test at screening and admission, non-lactating and of non-child bearing potential confirmed
4. Agree to use acceptable methods of contraception
5. Should not donate egg and sperm from the time of administration of treatment or study medication until 3 months following dose of study medication
6. Must be capable of understanding and complying with the requirements of the protocol and must have signed the informed consent form prior to undergoing any study-related procedures

Exclusion Criteria:

1. Male subjects with a female partner(s) who is (are) pregnant or lactating from the time of the administration of study medication
2. Has a clinically significant disease or any condition or disease that might affect drug absorption, distribution or excretion, e.g. gastrectomy, diarrhoea.
3. History of allergic reactions to artemisinin-based compounds, 4-aminoquinolines such as piperaquine or any other clinically relevant allergy to drugs or food.
4. Any clinically relevant history of cow's milk intolerance/allergy.
5. Any clinically significant abnormal laboratory, vital signs or other safety findings as determined by medical history, physical examination or other evaluations conducted at screening or on admission. Exception is PR, QTcB, QTcF, cardiac rhythm, liver function tests and haemoglobin that must be within the normal reference range at screening and on admission.
6. History or current evidence of any clinically relevant cardiovascular, pulmonary, hepatic, renal, gastrointestinal (excluding appendectomy and cholecystectomy), haematological, endocrinological, immunological, metabolic, neurological, oncological, psychiatric, urological or other disease, or current infection
7. History of post-antibiotic colitis
8. Electrocardiogram abnormalities in the standard 12-lead (at screening) and/or 24-hour 5 lead Holter (at screening) which in the opinion of the Investigator is clinically relevant or will interfere with the analysis
9. A history of clinically significant electrocardiogram abnormalities, or any of the following abnormalities at screening or admission:

   * PR >200 msec
   * QRS complex >120 msec
   * QTcB or QTcF >450 msec or shortened QTcB or QTcF less than 340 msec for males and females or family history of long QT syndrome or sudden death
   * Any degree of heart block (such as first, second or third degree atrioventricular block, incomplete, full or intermittent bundle branch block)
   * Abnormal T wave morphology / prominent U waves
   * Potassium levels out of the normal range at screening and prior to dosing
10. Positive results in any of the serology tests for Hepatitis B Surface Antigen, anti Hepatitis core antibody, Hepatitis C antibodies, and Human Immunodeficiency Virus 1 and 2 antibodies
11. Confirmed positive results from urine drug screen (amphetamines, benzodiazepines, cocaine, cannabinoids, opiates, barbiturates, and methadone) or from the alcohol breath test at screening and admission
12. History or clinical evidence of alcohol abuse, or any recreational drug abuse within the 2 years prior to screening
13. Mentally handicapped
14. Participation in a drug trial within 90 days prior to drug administration
15. Use of ANY prescription or over the counter medications, within 3 weeks of study drug administration, or vitamins or herbal supplements within 2 week of administration of the drug administration of study drug (or at least 5 half-lives of the compound whichever period is the longer), unless prior approval is granted by both the Investigator and Sponsor. Excluded from this list is intermittent use of paracetamol at up to 2g/day.
16. Use moderate or strong inhibitors and/or inducers of cytochrome CYP450 within 4 weeks prior to the planned drug administration (or at least 5 half-lives of the compound whichever period is the longer)
17. Subjects have veins unsuitable for intravenous puncture or cannulation on either arm (e.g. veins that are difficult to locate, access or puncture veins with a tendency to rupture during or after puncture)
18. Blood liver function tests not in the normal range at screening and on admission
19. Haemoglobin is less than the lower limit of the reference range at screening and on admission.
20. Donation of more than 500mL blood within 90 days prior to drug administration
21. Subjects must be non-smokers for at least 3 months prior to screening Note: "Tobacco use" includes smoking and the use of snuff and chewing tobacco, and other nicotine or nicotine containing products
22. Any consumption of grapefruit, Seville oranges, wild grapes, black mulberries, pomegranates in the form of fruit juice, marmalade or as a raw fruit within 7 days prior to dosing of study drug and throughout the study. Any circumstances or conditions, which, in the opinion of the investigator may affect full participation in the trial or compliance with the protocol
23. Legal incapacity or limited legal capacity at screening
24. Vegetarians, vegans or any dietary restrictions conflicting with the study standardised menus

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Lorch, MD FRCA FFPM, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Richmond Pharmacology Limited, Croyden, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment A: PQP 1440mg & OZ439+TPGS 800mg: PQP tablets 1440mg and OZ439+TPGS 800mg co-administered as a single oral dose fasted.
- Treatment B: PQP 960mg & OZ439+TPGS 800mg: PQP tablets 960mg and OZ439+TPGS 800mg co-administered as a single oral dose fasted.
- Treatment C - PQP 1440mg & OZ439 PIB 800mg: PQP Tablets 1440 mg and OZ439 PIB 800mg + full fat cow's milk
Period: Overall Study
Arm/Group | Treatment A: PQP 1440mg & OZ439+TPGS 800mg | Treatment B: PQP 960mg & OZ439+TPGS 800mg | Treatment C - PQP 1440mg & OZ439 PIB 800mg
Started | 8 | 8 | 8
Completed | 8 | 7 | 8
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All 24 subjects who had received at least one treatment of randomised study medication and for whom any post-treatment data was available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A: PQP 1440mg & OZ439+TPGS 800mg | Treatment B: PQP 960mg & OZ439+TPGS 800mg | Treatment C - PQP 1440mg & OZ439 PIB 800mg | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (13.06) | 30.1 (6.33) | 30.1 (5.79) | 31.3 (8.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1
  Male | 7 | 8 | 8 | 23
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: OZ439 Cmax
Description: OZ439 maximum concentration observed
Time Frame: Day 1 pre-dose and post-dose at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16 and 24 hours(Day 2), and, 48 (Day 3), 72 (Day 4), 96 (Day 5),168 (Day 8), Day 11, Day 15, Day 29 and Day 43
Population: Pharmacokinetic parameters were evaluated using all available concentration data from all 24 subjects who had received at least one treatment of randomised study medication.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: PQP 1440mg & OZ439+TPGS 800mg | Treatment B: PQP 960mg & OZ439+TPGS 800mg | Treatment C - PQP 1440mg & OZ439 PIB 800mg
Number analyzed (Participants) | 8 | 8 | 8
ng/mL | 1540 (26.0) | 1360 (33.8) | 1610 (37.2)

2. Primary Outcome: OZ439 AUC0-inf
Description: Area under the OZ439 plasma concentration time curve from time zero to time infinity using observed values.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: PQP 1440mg & OZ439+TPGS 800mg | Treatment B: PQP 960mg & OZ439+TPGS 800mg | Treatment C - PQP 1440mg & OZ439 PIB 800mg
Number analyzed (Participants) | 8 | 8 | 8
ng*h/mL | 17500 (27.9) | 16000 (24.7) | 18600 (45.4)

3. Secondary Outcome: Piperaquine Cmax
Description: Piperaquine maximum concentration observed
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: PQP 1440mg & OZ439+TPGS 800mg | Treatment B: PQP 960mg & OZ439+TPGS 800mg | Treatment C - PQP 1440mg & OZ439 PIB 800mg
Number analyzed (Participants) | 8 | 8 | 8
ng/mL | 202 (37.6) | 122 (42.1) | 630 (54.4)

4. Secondary Outcome: Piperaquine AUC0-inf
Description: Area under the Piperaquine plasma concentration time curve from time zero to time infinity using observed values.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: PQP 1440mg & OZ439+TPGS 800mg | Treatment B: PQP 960mg & OZ439+TPGS 800mg | Treatment C - PQP 1440mg & OZ439 PIB 800mg
Number analyzed (Participants) | 8 | 8 | 8
ng*h/mL | 17200 (29.5) | 13400 (23.1) | 29700 (48.0)

ADVERSE EVENTS:
Time Frame: Up to Day 43 post-dose.
Arm/Group | Treatment A: PQP 1440mg & OZ439+TPGS 800mg | Treatment B: PQP 960mg & OZ439+TPGS 800mg | Treatment C - PQP 1440mg & OZ439 PIB 800mg
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 6/8 | 4/8 | 5/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A: PQP 1440mg & OZ439+TPGS 800mg (N=8) | Treatment B: PQP 960mg & OZ439+TPGS 800mg (N=8) | Treatment C - PQP 1440mg & OZ439 PIB 800mg (N=8)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal Allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Change of bowel habit (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 3 (3) | 1 (1) | 3 (3)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After completion of the study, the Investigator may prepare a joint publication with the Sponsor. The Investigator must undertake not to submit any part of the individual data from this protocol for publication without prior consent of the Sponsor at a mutually agreed time.